CLINICAL TRIAL: NCT04946851
Title: Addictions Neuroclinical Assessment
Brief Title: Addictions Neuroclinical Assessment (ANA)
Status: Enrolling by invitation | Type: Observational
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000406; 000406-AA
Record Dates: First submitted 2021-06-30; First posted 2021-07-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-05-20

CONDITIONS: Normal Physiology; Alcohol Use Disorder
Keywords: Executive Function; Incentive Salience; Negative emotionality; Neurobiology; Alcohol Use Disorder; Natural History
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-treatment-seeking individuals: Participants across the spectrum of drinking (from non-drinkers to heavy drinkers) who are not interested in treatment for alcohol use disorder
- treatment-seeking individuals with alcohol use disorder: Volunteers with an AUD diagnosis who are seeking treatment for the condition

SUMMARY:
Background:

Alcohol use disorder (AUD) is a major public health problem. In the U.S., 16 to 18 million adults have an AUD. Researchers want to test an assessment tool called the ANA. It uses self-report and behavioral measures to assess 3 neuroscience domains of addiction. They hope to better understand, manage, prevent, and treat AUD.

Objective:

To learn how people s brains function related to their drinking.

Eligibility:

People ages 18 years and older who have enrolled in NIAAA natural history study 14-AA-0181.

Design:

Participants will complete surveys and tasks on a computer. The surveys and tasks assess a range of aspects of thinking and making decisions. The surveys and tasks also assess behaviors and feelings about alcohol and other rewards, and negative emotions. Participants will spend 90 minutes on the computer. Then they will take a break. In total, they will spend 4 blocks of time on the computer. Each block will last 90 minutes. They will take a break in between each block of time. They can take more breaks if needed.

Outpatient participants and healthy volunteers will complete this study in 1 visit. It will last about 6 hours. A second visit may be scheduled if needed. Outpatient participants will take a breath alcohol test. If their test is positive, their visit may be rescheduled or they may be withdrawn from the study.

Inpatient participants will complete this study over several days.

Data collected from participants in this study may be combined and analyzed with their data from NIAAA study 14-AA-0181 and/or NIAAA imaging study 14-AA-0080....

DETAILED DESCRIPTION:
Study Description:

This is a protocol examining a battery of assessments designed to study three neurofunctional domains relevant to alcohol use disorder (AUD), negative emotionality, incentive salience and executive function. The study will examine the relationships among the three ANA domains with the goal of identifying sub-types of AUD based on variation in the ANA domains.

Objectives:

Primary Objectives:

1. To examine the relationship between the three ANA domains

   (i.e. Negative Emotionality, Incentive Salience, Executive Function).
2. To identify the different subtypes of AUD based on variation in the ANA domains.

Secondary Objectives: None

Endpoints: Primary Endpoint: Latent factors of each of the ANA domains:

* Negative emotionality
* Incentive Salience
* Executive Function

Secondary Endpoints: None

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet both of the following criteria:

1. Participants must be > 18 years of age
2. Participants must have enrolled in the NIAAA Screening Protocol (14-AA-0181).

EXCLUSION CRITERIA:

There are no formal exclusionary criteria for this study. Based on enrollment criteria for the NIAAA Screening Protocol, individuals less than 18 years of age, or prisoners will not be enrolled in this study.

Outpatients will be tested for acute intoxication/impairment at the time of consent and study procedures using an alcohol breathalyzer and a clinical evaluation. Individuals with a positive breath alcohol concentration (BrAC), or those who are determined to be acutely intoxicated or impaired by the clinicians will be re-scheduled or withdrawn from the study.

In addition, individuals who are determined by the clinicians to be uncooperative or unable to provide consent, will not be invited to participate in this study. Individuals who report not being able to use a mouse and keyboard, or who are determined by the clinical research team to be unable to use a mouse and keyboard, will not be invited to participate in this study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population for this study includes adults across the spectrum of alcohol use who have been screened under the NIAAA screening protocol (14-AA-0181). This sample includes non-drinkers, light drinkers, non-treatment-seeking heavy drinkers, and treatment-seeking individuals with alcohol use disorder. Recruitment will be open to all participants from the NIAAA screening protocol.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2021-08-12 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
To examine the relationship between the three ANA domains (i.e. Negative Emotionality, Incentive Salience, Executive Function). | 1 visit
  Once the latent factors associated with each of the three ANA domains are identified, structural relationships between the latent factors can be modeled and described.
To identify the different subtypes of AUD based on variation in the ANA domains. | 1 visit
  Additionally, once the latent factors are identified, they can be used to categorize individuals into latent groups (AUD subtypes) based on the variation of their scores on each of the domains.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Diazgranados, M.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kwako LE, Schwandt ML, Ramchandani VA, Diazgranados N, Koob GF, Volkow ND, Blanco C, Goldman D. Neurofunctional Domains Derived From Deep Behavioral Phenotyping in Alcohol Use Disorder. Am J Psychiatry. 2019 Sep 1;176(9):744-753. doi: 10.1176/appi.ajp.2018.18030357. Epub 2019 Jan 4. PMID 30606047
- [Background] Kwako LE, Momenan R, Grodin EN, Litten RZ, Koob GF, Goldman D. Addictions Neuroclinical Assessment: A reverse translational approach. Neuropharmacology. 2017 Aug 1;122:254-264. doi: 10.1016/j.neuropharm.2017.03.006. Epub 2017 Mar 7. PMID 28283392
- [Background] Kwako LE, Momenan R, Litten RZ, Koob GF, Goldman D. Addictions Neuroclinical Assessment: A Neuroscience-Based Framework for Addictive Disorders. Biol Psychiatry. 2016 Aug 1;80(3):179-89. doi: 10.1016/j.biopsych.2015.10.024. Epub 2015 Nov 17. PMID 26772405
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000406-AA.html